CLINICAL TRIAL: NCT01981876
Title: Study of Esophageal Squamous Dysplasia Prevalence at Tenwek Hospital
Acronym: STEP
Status: Completed | Type: Observational
Sponsor: Tenwek Hospital (Other)
Collaborators: Kenyatta National Hospital (Other Government); Mayo Clinic (Other); AORTIC (Unknown)
Responsible Party: Sponsor
Other Study IDs: P172/06/2010
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Esophageal Dysplasia
Keywords: Dysplasia; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine specimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Esophageal squamous cell cancer (ESCC) is common in the developing world, and is the leading cancer diagnosis at Tenwek Hospital in southwestern Kenya. The investigators long-term goal is to understand the pathogenesis and risk factors for ESCC in Kenya, and to establish effective screening and prevention programs. The investigators hypothesize that asymptomatic esophageal squamous dysplasia (ESD) is common in their region, and the current protocol is designed to determine the prevalence of ESD in residents of southwestern Kenya.

DETAILED DESCRIPTION:
The prevalence of esophageal squamous dysplasia will be determined after evaluating pathology reports from unstained lesions and normal biopsies after staining with Lugol's iodine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* No dysphagia (subjects will be asked "do you have trouble swallowing food or water? Do they get stuck inside after you swallow?" in their primary language

Exclusion Criteria:

* Cardiac, respiratory, or metabolic disease that would increase the risk of endoscopy: history of myocardial infarction, arrhythmias, chronic obstructive pulmonary disease, diabetes, allergy to lidocaine.
* Unable or unwilling to provide informed consent.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Asymptomatic subjects residing within a 50 kilometer radius of Tenwek Hospital
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage rate of subjects with Esophageal Squamous dysplasia calculated as Prevalence | 2 years

SECONDARY OUTCOMES:
percentage of subjects with severe esophageal squamous dysplasia calculated as a prevalence | 2 years
percentage of subjects with moderate esophageal squamous dysplasia calculated as a prevalence | 2 years
percentage of subjects with mild esophageal squamous dysplasia calculated as a prevalence | 2 years

OTHER OUTCOMES:
Distribution of dysplasia rate by age | 2 years
  An analysis of dysplasia rates in each percentile age group
Distribution of unstained lesions on the esophagus by anatomic location | 2 years
  Distribution of unstained lesions on the esophagus based on their anatomic location after staining with lugol's iodine
Distribution of dysplasia rate by gender | 2 years
  Distribution of dysplasia rates by sex of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Mwachiro, MBChB, Principal Investigator — Tenwek Hospital; Russ E White, MD, Study Chair — Tenwek Hospital
Locations (1):
- Tenwek Hospital, Bomet, Riftvalley, Kenya